CLINICAL TRIAL: NCT01651858
Title: Nurigra Chewable Tablet in Healthy Adult Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: DW_SDF001
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nurigra Chewable tablet (Experimental)
  Interventions: Drug: Nurigra Chewable tablet
- Viagra (Active Comparator)
  Interventions: Drug: Nurigra Chewable tablet

INTERVENTIONS:
Drug: Nurigra Chewable tablet — 1 tablet of 100mg, once a day

SUMMARY:
The purpose of this study is to evaluate pharmacokinetics of sildenafil citrate in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and male subjects aged 20 to 45 years
* A Subject who was judged to be healthy by the investigator to participate in this study based on screening results (according to standard reference index updated recently)
* A subject who provided written informed consent to participate in this study and cooperative with regard to compliance with study related constraints.

Exclusion Criteria:

* A subject with sign or symptoms or previously diagnosed disease of liver

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2012-02; Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
to Assess Pharmacokinetics | 24h after drug administration
  AUC and Cmax in plasma

SECONDARY OUTCOMES:
to Assess Safety | 24h after administration
  Adverse events, Physical exam, Vital sign, Laboratory, 12-lead-ECG